CLINICAL TRIAL: NCT00332020
Title: RECORD 2 Study: REgulation of Coagulation in ORthopedic Surgery to Prevent DVT and PE, Controlled, Double-blind, Randomized Study of BAY 59-7939 in the Extended Prevention of VTE in Patients Undergoing Elective Hip Replacement.
Brief Title: Regulation of Coagulation in Orthopedic Surgery to Prevent DVT and PE, a Controlled, Double-blind, Randomized Study of BAY 59-7939 in the Extended Prevention of VTE in Patients Undergoing Elective Total Hip Replacement
Acronym: RECORD 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11357; 2005-004691-20 (EudraCT Number)
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Prevention; Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Rivaroxaban (BAY59-7939)
- Arm 2 (Active Comparator)
  Interventions: Drug: Enoxaparin

INTERVENTIONS:
Drug: Rivaroxaban (BAY59-7939) — 10 mg rivaroxaban (tablet) once daily administered for 35 +/- 4 days
  Arms: Arm 1
Drug: Enoxaparin — 40 mg enoxaparin syringe administered for 12 +/- 2 days
  Arms: Arm 2

SUMMARY:
The purpose of this study is to assess if 10 mg BAY 59-7939, taken once daily as a tablet, is safe and can help prevent blood clots forming after a hip replacement operation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 years or above
* Patients scheduled for elective total hip replacement

Exclusion Criteria:

* Planned, staged total bilateral hip replacement
* Active bleeding or high risk of bleeding contraindicating treatment with low molecular weight heparin
* Contraindication listed in the labeling or conditions precluding patient treatment with enoxaparin
* Conditions prohibiting bilateral venography (e.g. amputation of one leg, allergy to contrast media)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2457 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Composite endpoint of total VTE i.e.: Any DVT (proximal and/or distal), Non fatal PE, Death of all causes | Treatment period: up to day 35+/-6

SECONDARY OUTCOMES:
Incidence of the composite endpoint comprising proximal DVT, non-fatal PE and VTE- related death (major VTE) | Treatment period: up to day 35+/-6
Incidence of symptomatic VTE (DVT, PE) | Treatment period: up to day 35+/-6
Incidence of DVT (total, proximal, distal) | Treatment period: up to day 35+/-6
Incidence of symptomatic VTE during follow-up | Follow-up period: following 35+/-6 days
The composite endpoint comprising major VTE and treatment-emergent major bleeding | For major VTE, treatment period: up to Day 35+/-6 ; for major bleeding, from first dose of double-blind study medication to up to two days after last dose of double-blind study medication
Incidence of the composite endpoint that results from the primary endpoint by substituting VTE related death for all death | Treatment period: up to day 35+/-6
Incidence of the composite endpoint that results from major VTE by substituting all cause mortality for VTE-related death | Treatment period: up to day 35+/-6
Treatment-emergent major bleedings | From first dose of double-blind study medication to up to two days after last dose of double-blind study medication

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (109):
- United States (5):
  - Birmingham, Alabama
  - Denver, Colorado
  - Bay Pines, Florida
  - Miami, Florida
  - Oklahoma City, Oklahoma
- Australia (6):
  - Canberra, Australian Capital Territory
  - Lismore, New South Wales
  - Sydney, New South Wales
  - Southport, Queensland
  - Geelong, Victoria
  - Melbourne, Victoria
- Brazil (7):
  - Belo Horizonte, Minas Gerais
  - Curitiba, Paraná
  - Passo Fundo, Rio Grande do Sul
  - Batatais, São Paulo
  - Marília, São Paulo
  - São Paulo, São Paulo
  - Rio de Janeiro
- Canada (9):
  - Red Deer, Alberta
  - Penticton, British Columbia
  - Winnipeg, Manitoba
  - Saint John, New Brunswick
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Thunder Bay, Ontario
  - Windsor, Ontario
- China (6):
  - Guangzhou, Guangdong
  - Jinan, Shandong
  - Qingdao, Shandong
  - Xi’an, Shanxi
  - Beijing
  - Shanghai
- Colombia (4):
  - Barranquilla
  - Bogotá
  - Cali
  - Medellín
- Denmark (8):
  - Copenhagen
  - Frederiksberg
  - Glostrup Municipality
  - Herlev
  - Holbæk
  - Hvidovre
  - Silkeborg
  - Viborg
- Estonia (2):
  - Tallinn
  - Tartu
- India (6):
  - Hyderabad, Andhra Pradesh
  - Secundrabad, Andhra Pradesh
  - Bangalore, Bangalore
  - Ludhiana, Punjab
  - Bangalore
  - Mumbai
- Indonesia (2):
  - Surabaya, Surabaya
  - Bandung, West Java
- Italy (7):
  - Genova
  - Lecco
  - Modena
  - Napoli
  - Parma
  - Siena
  - Udine
- Latvia (2):
  - Liepāja
  - Riga
- Lithuania (4):
  - Kaunas
  - Klaipėda
  - Panevezys
  - Šiauliai
- Mexico (2):
  - Chihuahua, Chih., Chihuahua
  - Guadalajara, Jalisco
- Auckland, New Zealand
- Norway (4):
  - Kongsvinger
  - Namsos
  - Oslo
  - Tynset
- Peru (3):
  - Callao
  - Lima
  - Lima Cercado
- Portugal (4):
  - Lisbon, Lisbon District
  - Setúbal, Setúbal District
  - Torres Vedras, Torres Vedras
  - Porto
- South Africa (5):
  - Bloemfontein, Freestate
  - Johannesburg, Gauteng
  - Randburg, Gauteng
  - Newcastle, KwaZulu-Natal
  - Cape Town, Western Cape
- South Korea (3):
  - Kyunggido, Kyunggido
  - Daegu
  - Seoul
- Sweden (9):
  - Falköping
  - Hässleholm
  - Kungälv
  - Lidköping
  - Örebro
  - Stockholm
  - Sundsvall
  - Varberg
  - Vaxjo
- Taiwan (2):
  - Kaohsiung City
  - Taoyuan District
- United Kingdom (8):
  - Chesterfield, Derbyshire
  - Dumfries, Dumfries and Galloway
  - Kirkcaldy, Fife
  - London, Greater London
  - Liverpool, Merseyside
  - Great Yarmouth, Norfolk
  - Northampton, Northamptonshire
  - Epsom, Surrey

REFERENCES:
- [Derived] Kakkar AK, Brenner B, Dahl OE, Eriksson BI, Mouret P, Muntz J, Soglian AG, Pap AF, Misselwitz F, Haas S; RECORD2 Investigators. Extended duration rivaroxaban versus short-term enoxaparin for the prevention of venous thromboembolism after total hip arthroplasty: a double-blind, randomised controlled trial. Lancet. 2008 Jul 5;372(9632):31-9. doi: 10.1016/S0140-6736(08)60880-6. Epub 2008 Jun 24. PMID 18582928
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/